CLINICAL TRIAL: NCT06284681
Title: Weight-focused vs. Weight-neutral Adaptive Biobehavioral Strategies for Improving Metabolic Health in Black Adults With Stage 1 Obesity: A Pilot Sequential Multiple Assignment Randomized Trial
Brief Title: Weight Inclusive and Adaptive Strategies to Enhance Cardiometabolic Health in Black Adults
Acronym: WISE Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Drew Sayer, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-300012557; 3P50MD017338-03S1 (NIH)
Record Dates: First submitted 2024-02-06; First posted 2024-02-29 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Obesity; Prehypertension; Hypertension; PreDiabetes; Type 2 Diabetes; Dyslipidemia
MeSH Terms: conditions — Obesity; Prehypertension; Hypertension; Prediabetic State; Diabetes Mellitus, Type 2; Dyslipidemias

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Weight-Focused Health Coaching with Intensified Lifestyle Approach for Nonresponders (Experimental): Participants will start with weight-focused health coaching for 7 weeks and individuals achieving <3% weight loss will be given a 4-month membership to the YMCA and enrolled in group fitness classes.
  Interventions: Behavioral: Weight-focused health coaching; Behavioral: Intensify lifestyle approach
- Weight-Neutral Health Coaching with Intensified Lifestyle Approach for Nonresponders (Experimental): Participants will start with weight-neutral health coaching for 7 weeks and individuals achieving <150 minutes of moderate physical activity will be given a 4-month membership to the YMCA and enrolled in group fitness classes.
  Interventions: Behavioral: Weight-neutral health coaching; Behavioral: Intensify lifestyle approach
- Weight-Focused Health Coaching with Enhanced Medical Management (Experimental): Participants will start with weight-focused health coaching for 7 weeks and individuals achieving <3% weight loss will meet with their primary care provider and health coach to consider additional or revised medication plans to address their weight and weight-related chronic conditions.
  Interventions: Behavioral: Weight-focused health coaching; Other: Augment with enhanced medical management
- Weight-Neutral Health Coaching with Enhanced Medical Management (Experimental): Participants will start with weight-neutral health coaching for 7 weeks and individuals achieving <150 minutes of moderate physical activity will meet with their primary care provider and health coach to consider additional or revised medication plans to address their weight and weight-related chronic conditions.
  Interventions: Behavioral: Weight-neutral health coaching; Other: Augment with enhanced medical management

INTERVENTIONS:
Behavioral: Weight-focused health coaching — Following the definition of structured lifestyle interventions within the current obesity clinical practice guidelines, the weight-focused health coaching intervention will be delivered as a multi-component behavior change intervention intended to produce clinically-important weight loss through consuming a healthy, energy-restricted diet and increasing physical activity.
  Arms: Weight-Focused Health Coaching with Enhanced Medical Management; Weight-Focused Health Coaching with Intensified Lifestyle Approach for Nonresponders
Behavioral: Weight-neutral health coaching — Dietary and physical activity prescriptions for the weight-neutral health coaching intervention will be similar to the weight-focused intervention except the diet prescription will be designed to fully meet daily estimated energy requirements rather than creating a negative energy balance and producing weight loss. Health coaches will not emphasize changes in body weight as an explicit goal or as a mediator of improved cardiometabolic health. Rather, health coaches will emphasize achieving diet and exercise behavioral goals as a direct means to improving cardiometabolic health independently of changes in body weight.
  Arms: Weight-Neutral Health Coaching with Enhanced Medical Management; Weight-Neutral Health Coaching with Intensified Lifestyle Approach for Nonresponders
Behavioral: Intensify lifestyle approach — Participants identified as non-responders to initial health coaching interventions may be re-randomized to receive a 4-month membership to the local YMCA and health coaches will assist participants in identifying and enrolling in at least 2 weekly group fitness classes at the YMCA.
  Arms: Weight-Focused Health Coaching with Intensified Lifestyle Approach for Nonresponders; Weight-Neutral Health Coaching with Intensified Lifestyle Approach for Nonresponders
Other: Augment with enhanced medical management — Participants identified as non-responders to initial health coaching interventions may be re-randomized to meet with the primary care provider and health coach to consider additional or revised medication plans to address their weight and weight-related chronic conditions.
  Arms: Weight-Focused Health Coaching with Enhanced Medical Management; Weight-Neutral Health Coaching with Enhanced Medical Management

SUMMARY:
The proposed 6-month pilot Sequential Multiple Assignment Randomize Trial (SMART) has two aims. The first and primary aim is to determine the feasibility of conducting a full-scale SMART to compare weight-focused (i.e., weight loss) and weight-neutral (i.e., weight loss is not an explicit goal) adaptive biobehavioral interventions for improving cardiometabolic health in Black adults with overweight or obesity (BMI ≥27 kg/m2) plus at least one weight-related cardiometabolic condition (high blood pressure, prediabetes or diabetes, and/or high cholesterol). Biobehavioral interventions are treatment strategies that combine lifestyle-based behavioral interventions such as eating a healthy diet and exercise with medications. In this study, participants will be randomly assigned to receive either weight-focused or weight-neutral health coaching for 7 weeks. At week 8, participants will be identified as either "responders" or "nonresponders" to the initial interventions. The threshold for response in the weight-focused condition is greater than or equal to 3% weight loss. The threshold for response in the weight-neutral condition is engaging in greater than or equal to 150 minutes of moderate physical activity for the 7 days prior to the week 8 study visit. Responders to the initial interventions will continue with health coaching on a biweekly basis for weeks 9-26 of the intervention. Nonresponders will be re-randomized to either intensify the lifestyle-based intervention by receiving a membership to the YMCA and enrolling in group fitness classes or augmenting the health coaching with enhanced medical management in partnership with their established primary care provider. The second aim is to use clinical data from the pilot SMART to estimate treatment effects and the between-person variability in these effects. Because this is a pilot study, these estimates will not be used to make comparisons or draw conclusions on the comparative effectiveness of intervention conditions. Rather, these data will be used to generate preliminary effect sizes that can be used to estimate the sample size required for a full-scale trial. Clinical trial feasibility data will be collected on an ongoing basis throughout the study and clinical data will be collected prior to initiating the intervention (baseline) and at week 8 (response visit) and week 26 (post-intervention visit).

ELIGIBILITY:
Inclusion Criteria:

Black or African American Race

* ≥18 years
* BMI ≥27 kg/m2 plus a diagnostic history of 1 or more of the following:

  * Prehypertension or hypertension
  * Prediabetes or type 2 diabetes
  * Dyslipidemia
* Has a primary care provider who is willing to participate in enhanced medical management condition as needed
* Access and ability to use a device with reliable internet connectivity
* Able to converse and read English
* Willingness to enroll in any possible intervention conditions
* Willingness to engage in post-intervention focus group

Exclusion Criteria:

* Presence of any condition precluding engagement in the prescribed diet or exercise interventions
* Currently engaged in a structured lifestyle-based or weight loss intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | baseline
  Time required to meet recruitment goal
Retention rate | week 26
  Number and proportion of participants completing the study
Response/Non-response rate to initial interventions | week 8
  The proportion of participants meeting pre-specified response criteria initial interventions
Attendance to health coaching sessions | week 26
  Number and proportion of health coaching sessions attended attendance
Treatment Credibility and Expectancy Questionnaire (CEQ) | baseline
  The CEQ measures how much the participant believes in the rationale for the study treatments and how much they expect the treatments to improve their health.
Treatment Credibility and Expectancy Questionnaire (CEQ) | week 8
  The CEQ measures how much the participant believes in the rationale for the study treatments and how much they expect the treatments to improve their health.
Treatment Preference | baseline
  Measures the participant's preference for different treatments used in the study.
Treatment Preference | week 8
  Measures the participant's preference for different treatments used in the study.
Family medicine clinic capacity for research | week 26
  Measurement of family medicine clinic capacity for research
Study visit duration | week 26
  Measurement of study visit duration
Time required for surveys completion | week 26
  Measurement of time required for participants to complete the survey packet completion
Response to weight-focused health coaching | Week 8
  Weight loss measured using family medicine clinic. scale. Greater than or equal to 3 percent weight loss is the threshold for "response" for the weight focused condition.
Response to weight-neutral health coaching measurement | Week 8
  Physical activity measured accelerometry (activPAL4). Greater than or equal to 150 weekly minutes of physical activity is the threshold for response for the weight-neutral condition.

SECONDARY OUTCOMES:
Change in blood pressure | Week 26
  Measured by mercury sphygmomanometer
Change in glucose | Week 26
  Fasting blood draw
Change in insulin | Week 26
  Fasting blood draw
Change in insulin sensitivity | Week 26
  Measured by the quantitative insulin sensitivity check index (QUICKI). QUICKI is derived from measures of fasting insulin and fasting glucose, and a QUICKI score below 0.357 indicates low insulin sensitivity.
Change in HbA1c | Week 26
  Fasting blood draw
Change in total cholesterol | Week 26
  Fasting blood draw
Change in LDL-cholesterol | Week 26
  Fasting blood draw
Change in HDL-cholesterol | Week 26
  Fasting blood draw
Change in triglycerides | Week 26
  Fasting blood draw
Change in Metabolic Syndrome Severity Score | Week 26
  Metabolic Syndrome Severity Scores below zero indicate a lower degree of metabolic syndrome compared to the average adult, scores near zero indicate an average degree of metabolic syndrome, and scores above zero indicate an above average degree of metabolic syndrome and future disease risk.

OTHER OUTCOMES:
Change in blood pressure | Week 8
  Measured by mercury sphygmomanometer
Change in glucose | Week 8
  Fasting blood draw
Change in insulin | Week 8
  Fasting blood draw
Change in HbA1c | Week 8
  Fasting blood draw
Change in total cholesterol | Week 8
  Fasting blood draw
Change in LDL-cholesterol | Week 8
  Fasting blood draw
Change in HDL-cholesterol | Week 8
  Fasting blood draw
Change in triglycerides | Week 8
  Fasting blood draw
Change in body weight | Week 26
  Measured using family medicine clinic scale
Change in physical activity | Week 26
  Measured accelerometry (activPAL 4)
Change in fat mass | Week 8
  Measured by bioelectrical impedance (InBody S10)
Change in fat mass | Week 26
  Measured by bioelectrical impedance (InBody S10)
Change in lean mass | Week 8
  Measured by bioelectrical impedance (InBody S10)
Change in lean mass | Week 26
  Measured by bioelectrical impedance (InBody S10)
Change in waist circumference | Week 8
  Measured by Gulick tape
Change in waist circumference | Week 26
  Measured by Gulick tape
Dietary intake measurement | Week 8
  Measured by 7-day food record on ASA24
Dietary intake measurement | Week 26
  Measured by 7-day food record on ASA24
Change in insulin sensitivity | Week 8
  Measured by the quantitative insulin sensitivity check index (QUICKI). QUICKI is derived from measures of fasting insulin and fasting glucose, and a QUICKI score below 0.357 indicates low insulin sensitivity.
Change in Metabolic Syndrome Severity Score | Week 8
  Metabolic Syndrome Severity Scores below zero indicate a lower degree of metabolic syndrome compared to the average adult, scores near zero indicate an average degree of metabolic syndrome, and scores above zero indicate an above average degree of metabolic syndrome and future disease risk.

CONTACTS AND LOCATIONS:
Overall Officials: Drew Sayer, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
Coded and cleaned scientific data - with all participant identifiers removed - from all time points and supporting information will be preserved and shared from resulting publication(s) to allow for validation and replication of the study. All participant identifying information (e.g., names, addresses, contact information) will be saved in a separate and secure file for future contact purposes via IRB-approved study personnel and protocols only. Study-related data will be available via PubMed Central following publication.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Study-related data and supporting information will be made freely-available on PubMed Central following publication.